CLINICAL TRIAL: NCT02167464
Title: Controlling Blood Pressure in Treatment Resistant Hypertension: A Pilot Study
Acronym: TRH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34HL105880 (NIH)
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2014-09

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The PI was blinded to clinic and group assignment when he conducted the final statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aldosterone Antagonist (Active Comparator): Prescribe an aldosterone antagonist such as Spironolactone 12.5-25 mg daily as a starting dose with a maximum recommended dose of 50 mg daily.
  Interventions: Drug: Aldosterone Antagonist
- Referral Hypertension specialist (Active Comparator): Referral to a hypertension specialist
  Interventions: Other: Referral Hypertension specialist
- Renin treatment-guided therapeutics (Active Comparator): Renin treatment-guided therapeutics. A treatment algorithm is provided to guide treatment based upon renin levels.
  Interventions: Drug: Renin treatment-guided Therapeutics
- Renin-guided therapeutics and referral (Active Comparator): Renin treatment-guided therapeutics and referral to hypertension specialist. Treatment based upon algorithm for treatment related to renin level in addition to referral to a hypertension specialist.
  Interventions: Drug: Renin treatment-guided Therapeutics; Other: Referral Hypertension specialist

INTERVENTIONS:
Drug: Renin treatment-guided Therapeutics — Patients are treated based upon their renin levels according to an approved algorithm.
  Arms: Renin treatment-guided therapeutics; Renin-guided therapeutics and referral
Other: Referral Hypertension specialist — Patients are referred to a hypertension specialist.
  Arms: Referral Hypertension specialist; Renin-guided therapeutics and referral
Drug: Aldosterone Antagonist — Spironolactone 12.5 - 25mg daily
  Arms: Aldosterone Antagonist

SUMMARY:
Comparative Effectiveness Research using an intent-to-treat approach in 8 clinics in South Carolina. The investigators will assess 4 efficacious approaches to controlling treatment-resistant hypertension (TRH): Aldosterone Antagonist, Referral to Hypertension Specialist, Renin Treatment-Guided Therapeutics, and combination of Hypertension Specialist and Renin Treatment-Guided Therapeutics. Patients with TRH are evaluated with the BpTRU device for an accurate and representative blood pressure measure on two occasions before entry into the study. Qualitative data from focus group discussions with practice staff, and patient surveys and interviews will provide contextual data to help explain why some interventions are more acceptable and successful than others.

DETAILED DESCRIPTION:
This is Comparative Effectiveness Research conducted in the real world of under-resourced primary care clinics in South Carolina. Four arms of the study are identified with two clinics/arm enrolling and following patients with TRH. The goal is to compare rates of BP control according to American Heart Association guidelines among the 4 arms, along with clinic and patient satisfaction with each approach.

Our hypothesis is that defining pathophysiological mechanisms (e.g. renin treatment-guided therapeutics) with or without referral to a hypertension specialist will improve blood pressure control over adding an aldosterone antagonist in eligible patients or just referring patients to a hypertension specialist.

This mixed-methods design captures medical and qualitative data to not only describe the outcome of blood pressure control, but to assess the impact of the four interventions on staff and patient satisfaction. Key patient data includes demographics, visits, blood pressure values, medications and laboratory data. Focus group discussions with practice staff before and after the study will document early attitudes toward each arm, any practice changes needed to implement each arm and any burdens of the intervention on the practice. Patient surveys and interviews will assess their satisfaction with each intervention along with their experiences in participating in this research project.

Treatment Resistant Hypertension is a common medical condition, and relatively ineffective treatment regimens are a significant contributing factor. The long-term goal is to establish practice and effective approaches for controlling blood pressure and reducing clinical complications and related health disparities.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Treatment Resistant Hypertension (TRH)
* On three or more hypertensive medications at therapeutic dose
* BpTRU measurement on two occasions of >135/85 without diabetes or chronic kidney disease or BP >125/75 if diabetes and/or chronic kidney disease.
* Mean of >10 BP readings of >135/85 mm mercury for those with no diabetes or chronic kidney disease
* Mean of >10 home BP readings of >125/75 mm mercury for those with diabetes and/or chronic kidney disease.

Exclusion Criteria:

* Less than 18 years of age
* Refuses or incompetent to provide consent
* BP controlled to goal in or outside the clinic
* Symptomatic or significant orthostatic hypotension (<20/10 on standing)
* Life-threatening or severe illness
* Currently on protocol
* Myocardial Infarction or stroke in the past 6 months
* Estimated Glomerular Filtration Rate <50 ml/1.7/min.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
blood pressure control | four months
  Blood pressure control will be assessed according to guidelines established by American Heart Association.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn A Laken, PhD, RN, Principal Investigator — Medical University of South Carolina
Locations (8):
- United States (8):
  - AnMed, Anderson, South Carolina
  - Beaufort Jasper Hampton Comprehensive Health, Beaufort, South Carolina
  - McLeod Family Medicine Center, Florence, South Carolina
  - Family Diagnostics, Holly Hill, South Carolina
  - Lovelace Family Medicine, Prosperity, South Carolina
  - Carolina Medical Affiliates, Spartanburg, South Carolina
  - Spartanburg Regional Health Services, Spartanburg, South Carolina
  - Palmetto Primary Care, Summerville, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified data file is available. Email Suparna Qanungo at MUSC.

REFERENCES:
- [Background] Laken MA, Dawson R, Engelman O, Lovelace O, Way C, Egan BM. Comparative effectiveness research in the "real" world: lessons learned in a study of treatment-resistant hypertension. J Am Soc Hypertens. 2013 Jan-Feb;7(1):95-101. doi: 10.1016/j.jash.2012.12.002. PMID 23321408
- [Result] Egan BM, Laken MA, Sutherland SE, Qanungo S, Fleming DO, Cook AG, Hester WH, Jones KW, Jebaily GC, Valainis GT, Way CF, Wright MB, Davis RA. Aldosterone Antagonists or Renin-Guided Therapy for Treatment-Resistant Hypertension: A Comparative Effectiveness Pilot Study in Primary Care. Am J Hypertens. 2016 Aug;29(8):976-83. doi: 10.1093/ajh/hpw016. Epub 2016 Apr 13. PMID 27076600